# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Evaluation of Approved and Investigational Contact Lenses

Protocol CR-5960

Version: 2.0

**Date:** 14 June 2017

Investigational Products: Senofilcon-based contact lens containing new-UV blocker

Key Words: senofilcon A, Subjective Performance, Fitting Characteristics, Dispensing, Daily

Wear

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP), ISO 14155, the Declaration of Helsinki, and all applicable regulatory requirements.

### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

### TABLE OF CONTENTS SPONSOR NAME AND ADDRESS......6 AUTHORIZED SIGNATURES 7 CHANGE HISTORY.....8 SYNOPSIS 9 1.1. 1.2. 1.3. 1.4. 15 Relevant Literature References and Prior Clinical Data Relevant to Proposed 2.1. 2.2. 2.3. General Characteristics 22 3 1 3.2. 3.3. Exclusion Criteria 23 3.4. Enrollment Strategy.......24 4. STUDY DESIGN AND RATIONALE 24 4.1. Description of Study Design 24 4.2. 43 5. TEST ARTICLE ALLOCATION AND MASKING .......25 5.1 5.2. 5.3.

| 6.1. Identity of Test Articles | 26 |
|-------------------------------------------------------|------|
| Table 1: Test Articles | 27 |
| 6.2. Ancillary Supplies/Products | 27 |
| Table 2: Ancillary Supplies | 27 |
| 6.3. Administration of Test Articles | 27 |
| 6.4. Packaging and Labeling | 27 |
| 6.5. Storage Conditions | 28 |
| 6.6. Collection and Storage of Samples | 28 |
| 6.7. Accountability of Test Articles | 28 |
| 7. STUDY EVALUATIONS | 29 |
| 7.1. Time and Event Schedule | 29 |
| Table 3: Time and Events | 29 |
| 7.2. Detailed Study Procedures | 30 |
| VISIT 1 | 30 |
| VISIT 2 | 34 |
| VISIT 3 | 36 |
| VISIT 4 | 40 |
| VISIT 5 | 44 |
| FINAL EVALUATION | 46 |
| 7.3. Unscheduled Visits | 46 |
| 7.4. Laboratory Procedures | 47 |
| 8. SUBJECTS COMPLETION/WITHDRAWAL | 48 |
| 8.1. Completion Criteria | 48 |
| 8.2. Withdrawal/Discontinuation from the Study | 48 |
| 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 49 |
| 10. DEVIATIONS FROM THE PROTOCOL | |
| 11. STUDY TERMINATION | 50 |
| 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 5050 |
| 13. ADVERSE EVENTS | 51 |
| 13.1. Definitions and Classifications | 51 |
| 13.2. Assessing Adverse Events | |
| 13.2.1 Causality Assessment | |
| 13.2.2 Severity Assessment | 54 |
| 13.3 Documentation and Follow-Up of Adverse Events | 55 |

| 13.4. | Reporting Adverse Events | 56 |
|---|---|---|
| 13. | .4.1 Reporting Adverse Events to Sponsor | . 56 |
| 13. | .4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities. | . 57 |
| 13.5. | Event of Special Interest | 57 |
| 13.6. | Reporting of Pregnancy | . 57 |
| 14. STA | ATISTICAL METHODS | . 58 |
| 14.1. | General Considerations | . 58 |
| 14.2. | Sample Size Justification. | . 58 |
| Table | 4: Historical Study Included in Sample Size Calculation | . 58 |
| Table | Descriptive Summary of CLUE Comfort, Unacceptable Lens Fit and Outdoor Performance Items Pooled across Historical Studies- 2-Week Follow-up evaluation | 59 |
| Table | e 6: Descriptive Summary of Slit Lamp Findings Pooled Across Historical Studies | . 59 |
| Table | e 7: Sample Size Estimates and Power Calculations for Primary Endpoints | . 60 |
| 14.3. | Analysis Populations | . 61 |
| 14.4. | Level of Statistical Significance | . 61 |
| 14.5. | Primary Analysis | . 61 |
| 14.6. | Secondary Analysis | . 66 |
| 14.7. | Other Exploratory Analyses | . 66 |
| 14.8. | Interim Analysis | . 69 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | . 69 |
| 14.10 | Procedure for Reporting Deviations from Statistical Plan | . 70 |
| 15. DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | . 70 |
| 15.1. | Electronic Case Report Form/Data Collection | . 70 |
| 15.2. | Subject Record | . 70 |
| 16. DA | TA MANAGEMENT | . 71 |
| | Access to Source Data/Document | |
| 16.2. | Confidentiality of Information | . 71 |
| 16.3. | Data Quality Assurance | . 71 |
| 17. MO | NITORING | . 72 |
| 18. ETI | HICAL AND REGULATORY ASPECTS | . 72 |
| 18.1. | Study-Specific Design Considerations | . 72 |
| 18.2. | Investigator Responsibility | . 73 |
| 18 3 | Independent Ethics Committee or Institutional Review Board (IEC/IRR) | 73 |

| 18.4. Informed Consent | 74 |
|---|---|
| 18.5. Privacy of Personal Data | 74 |
| 19. STUDY RECORD RETENTION | 75 |
| 20. FINANCIAL CONSIDERATIONS | 76 |
| 21. PUBLICATION | 76 |
| 22. REFERENCES | 77 |
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 78 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | 97 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APPENDIX D: CLINICAL TECHNICAL PROCEDURES | 101 |
| , LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS | |
| , EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 110 |
| , LENS FITTING CHARACTERISTICS | 115 |
| , SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | 122 |
| , FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDUR | E124 |
| , DETERMINATION OF DISTANCE SPHEROCYLINDRICAL | |
| REFRACTIONS | |
| , BIOMICROSCOPY SCALE | |
| , DISTANCE AND NEAR VISUAL ACUITY EVALUATION | |
| , DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDUR | |
| APPENDIX E: IRIS Color | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 154 |
| LISTING OF TABLES | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |
| Table 5: Descriptive Summary of CLUE Comfort, Unacceptable Lens Fit | |
| Outdoor Performance Items Pooled across Historical Studies- 2-Week Follow-up evaluat | |
| Table 6: Descriptive Summary of Slit Lamp Findings Pooled Across Historical Studies<br>Table 7: Sample Size Estimates and Power Calculations for Primary Endpoints | |
| LISTING OF FIGURES | |
| Figure 1: Study Flowchart | 1/ |

### PROTOCOL TITLE, NUMBER, VERSION

Title: Evaluation of Approved and Investigational Contact Lenses

Protocol Number: CR-5960

Version: 2.0

Date: 14 June 2017

### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway, Jacksonville, FL 32256

### MEDICAL MONITOR

Name: John R. Buch, O.D., M.S., F.A.A.O. Title: Principal Research Optometrist Address:

Email: jbuch@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155 and the Declaration of Helsinki.

| Author | See Electronic Signature Report | DATE |
|---|---|---|
| | Title: Principal Research Optometrist | |
| Clinical Operations<br>Manager | See Electronic Signature Report | |
| Manager | | DATE |
| | Title: Clinical Operations Manager | |
| Biostatistician | See Electronic Signature Report | |
| | Title: Biostatistician II | DATE |
| Biostatistician | | |
| Reviewer | See Electronic Signature Report | DATE |
| | Title: Manager of Biostatistics | |
| Reviewer | See Electronic Signature Report | DATE |
| | Title: Clinical Research Fellow | DITTE |
| Data Management | See Electronic Signature Report | |
| | Title: Clinical Project Manager, Data and | DATE |
| | Systems | |
| Approver | See Electronic Signature Report | DATE |
| | Title: Reusable Platform Lead | DATE |

### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section Number(s)<br>Affected | Date |
|---|---|---|---|
| 1.0 | | New protocol | 09 June 2017 |
| 2.0 | | Corrected grammatical errors in Patient Reported Outcomes (Study Questionnaire): Page 84 – added "your" to Item ID# MIN00246; pages 92 and 93 – added comma to Item ID#s PREF12 and PREF10. | |

### **SYNOPSIS**

| Protocol Title | Evaluation of Approved and Investigational Contact Lenses |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development Phase 2b |
| Trial Registration | This study will be registered on ClinicalTrials.gov after final product approval from the FDA. |
| Test Article(s) | Investigational Products: Senofilcon-based contact lens containing new-UV blocker (a.k.a. Test lens) |
| | Control Products: Commercial ACUVUE® OASYS® |
| Wear and Replacement<br>Schedules | Wear Schedule: daily wear (DW) |
| | Replacement Schedule: approximately 2 weeks |
| Objectives | The primary objective of this study is to demonstrate non-inferiority of the Test lens compared to the Control lens with respect to CLUE comfort, Slit Lamp Findings and Monocular logMAR Distance Visual Acuity. This study will also aim to show the Fit Acceptance rate is at least 90% in order to assess performance of the Test lens for eventual Design Validation and/or Claims studies. |
| Study Endpoints | Primary Endpoints: |
| | <ul> <li>Monocular logMAR distance visual acuity</li> <li>Biomicroscopy</li> <li>Fit acceptance rate</li> <li>Overall CLUE comfort</li> </ul> |
| | Secondary Endpoints: |
| | <ul><li>Overall CLUE vision</li><li>Overall CLUE handling</li></ul> |

| Study Design | This study is a randomized, 5-visit, partial subject-masked, 2×3 bilateral crossover, dispensing trial. The study lenses will be worn as daily wear (DW) for a period of 2 weeks each with one of the study lenses being worn twice. Each study lens is expected to be worn at least five (5) days per week for at least six (6) hours per day worn. There will be no washout period between study lenses. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations. |
|---|---|
| Sample Size | Approximately 130 eligible subjects will be enrolled and randomized into the study. Approximately 120 subjects are targeted to complete the study. A replacement subject may be enrolled if a subject discontinues from the study prematurely; the decision whether to enroll replacement subjects will be made by the joint agreement of the Investigator and Sponsor. |
| Study Duration | Subjects will wear the Test and control lenses for 2 weeks each in random order with one of the study lenses being worn twice for a total of 6 weeks per subject. The enrollment period will be 2 weeks, making the entire study approximately 8 weeks in duration. |
| Anticipated Study<br>Population | Approximately 130 subjects will be enrolled to ensure that at least 120 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of ≥18 and ≤49. |

### Eligibility Criteria Potential subjects must satisfy all of the following inclusion criteria to be enrolled in the study: (Inclusion Criteria) 1. The subject must read and sign the Informed Consent 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol. 3. Healthy adult males or females age $\geq$ 18 and $\leq$ 49 years of age with signed informed consent. presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. 4. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and -6.00D. 5. The subject's refractive cylinder must be $\leq 1.00D$ in each eve. 6. The subject must have visual acuity best correctable to 20/25+3 or better for each eye. 7. Subjects must own a wearable pair of spectacles. 8. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis. 9. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per 10. The subject must have normal eyes (i.e., no ocular medications or infections of any type). Eligibility Criteria Potential subjects who meet any of the following criteria will be excluded from participating in the study: (Exclusion Criteria) 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued). 2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis). 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g.

Accutane), oral tetracyclines, topical scopolamine, oral

- (e.g., Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
- 4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
- 5. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 6. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g.., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
- 7. Any known hypersensitivity or allergic reaction to Optifree®PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution
- 8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
- 9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
- 10. Toric, extended wear, monovision or multi-focal contact lens correction.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
- 13. History of binocular vision abnormality or strabismus.
- 14. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).


| | <del>,</del> |
|---|---|
| Disallowed Medications/Interventions | Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication |
| Measurements and Procedures | Monocular distance visual acuity on logMAR scale using ETDRS charts, physiological responses, fitting characteristics, individual performance metrics, CLUE comfort, vision and handling. |
| Microbiology or Other<br>Laboratory Testing | The optical bench will be used to measure the light transmission characteristics for all worn test lenses. The findings are for internal information only and will not be part of the final report. |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the control lens of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Opti-Free® PureMoist®, Preservative free rewetting drops/artificial tears |
| Principal Investigator(s)<br>and Study<br>Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

CTP Clinical Technical Procedure

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

logMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide

PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity UV Ultraviolet

HEV High energy visible PG Propylene glycol IPA Isopropyl alcohol

### 1. INTRODUCTION AND BACKGROUND

ACUVUE® OASYS® is manufactured with a UV-blocker that blocks at least 99% of UV-B radiation and at least 90% of UV-A radiation (i.e., Class 1 UV-blocking). The new UV-blocker in the Test lens extends these radiation-blocking capabilities.

### 1.1. Name and Descriptions of Investigational Products

Senofilcon-based contact lens containing a new-UV blocker.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigative product in this study is for correcting myopia and providing visual benefits in lighting situations where UV-A and/or High Energy Visible (HEV) light is present in the environment. During the study, each test article will be worn bilaterally in a daily wear modality for at least 6 hours per day and 5 days per week for approximately 2 weeks each. The subject will wear either the Test or Control article twice and the other study article once.

### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans.

### 1.4. Known Risks and Benefits to Human Subjects

and Informed Consent. The material safety testing/lens release criteria was determined based on the Risk Assessment.

### 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

The literature is absent of any articles pertaining to soft contact lenses containing the new type of UV-blocker. A list of relevant literature references pertaining to glare, eyestrain, and light filtering is provided:

- Agarwal, S., Goel, D., & Sharma, A. (2013). Evaluation of the factors which contribute to the ocular complaints in computer users. J Clin Diagn Res,7(2), 331-335.
- 2. Eperjesi, F., Fowler, C. W., & Evans, B. J. (2002). Do tinted lenses or filters improve visual performance in low vision? A review of the literature. Ophthalmic and Physiological Optics, 22(1), 68-77.
- Hickcox, K. S., Narendran, N., Bullough, J. D., & Freyssinier, J. P. (2013). Effect of different coloured luminous surrounds on LED discomfort glare perception. Lighting Research and Technology, 1477153512474450.


- 4. Leguire, L. E., & Suh, S. (1993). Effect of light filters on contrast sensitivity function in normal and retinal degeneration subjects. Ophthalmic and Physiological Optics, 13(2), 124-128.
- 5. Morse, R. S. (1985, October). Glare filter preference: influence of subjective and objective indices of glare, sharpness, brightness, contrast and color. In Proceedings of the Human Factors and Ergonomics Society Annual Meeting(Vol. 29, No. 8, pp. 782-786). SAGE Publications.
- 6. Pérez-Carrasco, M. J., Puell, M. C., Sánchez-Ramos, C., López-Castro, A., & Langa, A. (2005). Effect of a yellow filter on contrast sensitivity and disability glare after laser in situ keratomileusis under mesopic and photopic conditions. Journal of Refractive Surgery, 21(2), 158-165.
- 7. Sheedy, J. E., Hayes, J., & ENGLE, J. (2003). Is all asthenopia the same?. Optometry & Vision Science, 80(11), 732-739.
- 8. Steen, R., Whitaker, D., Elliott, D. B., & Wild, J. M. (1994). Age-related effects of glare on luminance and color contrast sensitivity. Optometry & Vision Science, 71(12), 792-796.
- 9. Vincent, A. J., Spierings, E. L., & Messinger, H. B. (1989). A controlled study of visual symptoms and eye strain factors in chronic headache. Headache: The Journal of Head and Face Pain, 29(8), 523-527.
- 10. Wilkins, A. J., & Evans, B. J. (2010). Visual stress, its treatment with spectral filters, and its relationship to visually induced motion sickness. Applied Ergonomics, 41(4), 509-515.

### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

### 2.1. Objectives

### Primary Objective

The primary objective of this study is to demonstrate non-inferiority of the Test lens compared to the Control lens with respect to CLUE comfort, Slit Lamp Findings and Distance Monocular logMAR Visual Acuity. This study will also aim to show that the Fit Acceptance rate is at least 90% for subjects wearing the Test lens.

### Secondary Objective

The secondary objective of this study is to demonstrate non-inferiority of the Test lens compare to the Control lens with respect to CLUE Overall quality of Vision and Handling.

### **Exploratory Objective**

This study also aims to explore the performance of Indoor, Outdoor and Driving performance using individual questionnaire items.

### 2.2. Endpoints

**Primary Endpoints** 

The primary endpoints are as follows:

### <u>Biomicroscopy</u>

Biomicroscopy will be assessed for each subject eye at all study visits (scheduled and unscheduled). The percentage of Grade 3 or higher slit lamp findings will be analyzed and will include corneal infiltrates.

### Distance Monocular Contact Lens Visual Acuity

Distance monocular contact lens visual performance (logMAR) is assessed for each subject eye at the 2-week follow-up evaluation.

### Fit Acceptance Rate

Acceptable lens fit will be assessed at all scheduled visits for each subject eye. Fit acceptance rate will be based on the lens fit acceptance of eyes wearing the Test lens only. Fit rates of the control lens will also be collected, but are not a primary endpoint.

### CLUE Overall Comfort

Overall comfort scores are assessed using the Contact Lens User Experience (CLUE) questionnaire at the two-week follow-up. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. (2016)<sup>1</sup>.

### Secondary Endpoints

The Secondary endpoints are as follows:

### CLUE Overall Quality of Vision and Handling

Overall Quality of vision and handling scores are assessed using the Contact Lens User Experience (CLUE) questionnaire at the 2-week follow-up. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response (2016)<sup>1</sup>.

### Other Observations

### Lens Preferences

Lens preferences will be assessed by patient reported outcome (PRO) questions regarding lens preference at the 2-week follow-up of the second wearing period. Subjects will be asked to choose for each preference item one of the following responses: Strongly Prefer the first lens, Prefer the first lens, no preference, prefer the second lens, strongly prefer the second lens. Lens preference questions consist of:






### Driving Performance

Driving performance will be assessed by two individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:



### **Indoor Performance**

Indoor performance will be assessed by three individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:



### **Outdoor Performance**

Outdoor performance will be assessed by four individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:



### 2.3. Hypotheses

### Primary Hypotheses

All primary and secondary hypotheses must be met in order to satisfy the objective the study.

| Primary Hypotheses | |
|---|---|
| Endpoint | Hypothesis |
| Monocular logMAR visual acuity | The Test lens will be non-inferior to the control lens with respect to Distance Monocular logMAR Visual Acuity at the 2-week follow-up evaluation. A non-inferiority margin of 0.05 logMAR and a superiority margin of 0 logMAR will be used. |
| Biomicroscopy | The Test lens will be non-inferior to the control lens with respect |

| | to the percentage of eyes with Grade 3 or higher Slit Lamp Findings (Biomicroscopy) across all follow-up visits (scheduled and unscheduled). A non-inferiority margin of 5% will be used. |
|---|---|
| Fit acceptance rate | The proportion of eyes with acceptable fit will be greater than 90% across all scheduled visits for all subjects wearing the Test lens. The fit acceptance rate of the control lens is not a primary endpoint. |
| Overall CLUE comfort | The Test lens will be non-inferior to the control lens with respect to CLUE Overall Comfort at the 2-week follow-up evaluation. A non-inferiority margin of -5 points will be used |

## Secondary Hypotheses

| Secondary Hypotheses | |
|---|---|
| Endpoint | Hypothesis |
| Overall CLUE Vision | The Test lens will be non-inferior to the control lens with respect to CLUE Overall quality of vision at the 2-week follow-up evaluation. A non-inferiority margin of -5 points will be used. |
| Overall CLUE handling | The Test lens will be non-inferior to the control with respect to CLUE Handling at the 2-week follow-up evaluation. A non-inferiority margin of -5 points will be used. |

## Other Hypotheses

| Other Observations | |
|---|---|
| Endpoint | Hypothesis |
| Lens Preferences | The Test lens will be superior to the control lens in all 5 of the following lens preference items at the 2-week follow-up evaluation of the second wearing period. |

| Other Observations | |
|---|---|
| Endpoint | Hypothesis |
| Indoor Performance<br>Measures | The Test lens will be superior to the control lens in at least 2 of the following 4 indoor performance measure(s) at the 2-week follow-up evaluation. |
| Driving Performance<br>Metrics | The Test lens will be non-inferior to the control lens in both of the following driving performance metrics at the 2-week follow-up evaluation. A cumulative odds ratio margin of 0.67 will be used. |
| Outdoor Performance<br>Measures | The Test lens will be superior to the control lens in at least 2 of the following 4 outdoor performance measure(s) at the 2-week follow-up evaluation. |

### Justification of Clinical Margins

- A 5 point increase in an average CLUE score translates into 10% shift in the distribution of scores for a population of soft contact lens wearers<sup>1</sup>.
- The cumulative odds ratio margin of 0.67 was selected since this corresponds to no more than a 10% difference in cumulative proportion between the Test and control groups.

### 3. TARGETED STUDY POPULATION

### 3.1. General Characteristics

Approximately 130 subjects will be enrolled to ensure that at least 120 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 and ≤49 years old. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear

the Test and Control contact lenses approximately 2 weeks each bilaterally on a daily wear (DW) basis, then wear either the Test or Control lens again for 2 weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The subject must read and sign the Informed Consent form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Healthy adult males or females age ≥18 and ≤49 years of age with signed informed consent. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
- 4. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and -6.00D.
- 5. The subject's refractive cylinder must be  $\leq$ 1.00D in each eye.
- 6. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
- 7. Subjects must own a wearable pair of spectacles.
- 8. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
- 9. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week
- 10. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
- 2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
- 4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.

- 5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 6. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g.., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
- 7. Any known hypersensitivity or allergic reaction to Optifree®PureMoist® multipurpose care solution or Eye-Cept® rewetting drop solution
- 8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
- 9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
- 10. Toric, extended wear, monovision or multi-focal contact lens correction.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
- 13. History of binocular vision abnormality or strabismus.
- 14. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).

### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

### 4. STUDY DESIGN AND RATIONALE

### 4.1. Description of Study Design

This study is a randomized, 5-visit, partial subject-masked,  $2\times3$  bilateral crossover, dispensing trial. Both study lenses will be worn as daily wear (DW) for a period of 2 weeks each, and each study lens is expected to be worn at least five (5) days per week for at least six (6) hours per day worn. There will be no washout period between study lenses.

### 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. This design was considered since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared a parallel study since fewer subjects are required to achieve the same pre-specified statistical power.

significant carryover effects were observed when assessing clinically relevant differences between the Test lens and a comparator while using a 2×2 crossover study design. Therefore this study utilizes a 3-period


by 2-treatment in order to estimate the true effect of the Test lens without any potential bias from the carry-over effect.

### 4.3. Enrollment Target and Study Duration

Approximately 130 subjects will be enrolled to ensure that at least 120 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 and ≤49 years old. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear the Test and Control contact lenses bilaterally approximately 2 weeks each on a daily wear (DW) basis, then wear either the Test or Control lens again for 2 weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

### 5. TEST ARTICLE ALLOCATION AND MASKING

### 5.1. Test Article Allocation

This is a multi-site, partially-subject masked (control lens only) and randomized study. The study lenses will be worn in a bilateral and random fashion using a 2 treatment by 3 period (2×3) crossover design.

Permuted block randomization will be used to minimize the potential for treatment imbalance. A block size of two (2) sequences will be utilized. A computer-generated randomization scheme will be used to randomly assign subjects to one of the two possible lens wear sequences (TEST/CONTROL/CONTROL or CONTROL/TEST/TEST). The random scheme will be generated using the PROC PLAN procedure from SAS Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment according to the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected

### 5.2. Masking

Complete masking is impossible due to the functioning nature of the Test lens. The control lens will be over-labeled to mask the identity since the control lens may be the subject's habitual lens by chance. Therefore the study is partially-subject masked (control lens only).

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the investigator may in an emergency contact the medical monitor. In the event the mask is broken, the sponsor must be notified before the

mask is broken. The date, time, and reason for the unmasking must be documented in the source document. The investigator is also advised not to reveal the study treatment assignment to the study site or sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

Use of the test articles will be randomized using a randomization scheme supplied by the study biostatistician.

If the test article is randomized, the order will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

### 5.3. Procedures for Maintaining and Breaking Randomization Codes

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Control | Test |
|---|---|---|
| Name | OASYS | ECL100 |
| Manufacturer | JJVC | JJVC |
| Compass Protocol(s) and/or Lot Number or | NA (Commercial | |
| Other Identifier | Product) | |
| Lens Material | senofilcon A | senofilcon A |
| Nominal Base Curve @ 22°C | 8.4 | 8.4 |
| Nominal Diameter @ 22°C | 14.0 | 14.0 |
| Nominal Distance Powers (D) | -1.00 to -6.00 in 0.25 | -1.00 to -6.00 in 0.25 |
| | steps | steps |
| Water Content (Optional) | 38 | 38 |
| Center Thickness (Optional) | 0.070 | 0.085 |
| Oxygen Permeability (Dk) | 103 | 103 |
| Modality in Current Study | Daily wear | Daily wear |
| Replacement Frequency | Single use | Single use |
| Packaging Form (vial, blister, etc.) | Sterile blister pack | Sterile blister pack |
| New-UV blocker concentration | NA | ~1.0% |

Approximately 75 lenses per sku will be made available based on the following factors: sample size, 2×3 design, bilateral wear, biweekly replacement, safety margin of 2x, and US distribution model for the range of lenses -1.00 through -6.00 D.

### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution 1 | Solution 2 |
|---|---|---|
| Solution Name / | Out Free R Down MaintR | Eye-Cept® |
| Description | Opti-Free® PureMoist® | Rewetting Drops |
| Lot Number or Other | Varies | Varies |
| Identifier | varies | Varies |
| Manufacturer | Alcon Laboratories, Fort Worth, TX | Optics Laboratories |
| Maximum | 0.001% polyquaternium-1, 0.0006% | NA |
| Preservative | myristamidopropyl dimethylamine | INA |

### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

### 6.4. Packaging and Labeling

The Test articles will be packaged in blisters as the primary packaging. The Control article will be over-labeled to mask the subject to the identity of the lens. The Test articles will be in


investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:

### US label A (for control lens over-label)



### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions and out of direct sunlight.

### 6.6. Collection and Storage of Samples

All worn study lenses will be collected from the subject, placed in labeled glass vials with Opti-Free<sup>®</sup> Puremoist<sup>®</sup>, and stored refrigerated or frozen until they are shipped back to the Sponsor. The lenses will be shipped in special containers to keep the lenses refrigerated.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the

clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will package and return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

: Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

### 7. STUDY EVALUATIONS

### 7.1. Time and Event Schedule

Table 3: Time and Events

| Procedure | Baseline | Trial Fit & Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 3, 4 | 2, 3, 4, 5 | PRN | 5 |
| Visit Window | - | - | 6-8 Days<br>13-15 Days | - | - |
| Informed consent | ✓ | - | - | - | - |
| Eligibility screening | ✓ | - | - | - | - |
| CLUE Baseline Questionnaire | ✓ | - | - | - | - |
| GSI Background Questionnaire | | | | | |
| Other Questionnaires | ✓ | - | ✓ | - | - |
| Subject demographics | ✓ | - | - | - | - |
| General health and medication history | <b>✓</b> | - | - | - | - |
| Subject's own contact lens information | ✓ | - | - | - | - |
| Habitual lens care | <b>√</b> | - | - | - | _ |
| Entrance visual acuity | <b>√</b> | - | - | - | - |
| Spherocylindrical refraction and BVA | ✓ | - | - | ✓ | <b>√</b> |
| Slit lamp biomicroscopy | ✓ | - | ✓ | ✓ | _ |
| Expanded Conjunctival Redness | ✓ | - | ✓ | ✓ | - |
| Expanded Corneal Staining | ✓ | - | ✓ | <b>√</b> | - |
| Trial fitting lens information | - | ✓ | - | - | - |
| Lens Damage | - | ✓ | - | - | - |
| Distance spherical over-<br>refraction | _ | ✓ | <b>√</b> | - | - |
| Lens modification | - | <b>√</b> | - | - | - |
| Visual acuity | - | <b>√</b> | ✓ | <b>√</b> | - |
| Lens fitting assessment | - | <b>√</b> | ✓ | * | - |

| Procedure | Baseline | Trial Fit &<br>Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 3, 4 | 2, 3, 4, 5 | PRN | 5 |
| Visit Window | - | - | 6-8 Days<br>13-15 Days | - | - |
| Lens wettability | - | ✓ | ✓ | * | - |
| Lens dispensing information and criteria | - | ✓ | - | - | 1 |
| Patient instructions | - | ✓ | - | - | - |
| Lens information | - | - | ✓ | ✓ | |
| Compliance | - | - | ✓ | ✓ | - |
| Wearing times | - | 1 | <b>✓</b> | ✓ | - |
| CLUE Follow-Up Questionnaire | - | ı | <b>✓</b> | * | - |
| GSI Product Performance<br>Questionnaire | - | - | ✓ | * | - |
| Symptoms | - | ✓ | ✓ | ✓ | - |
| Lens preference | - | - | V 2, 3, 4 | - | - |
| Surface characteristics | - | - | ✓ | * | - |
| Chief complaint, diagnosis, treatment | - | - | - | ✓ | - |
| * if wearing study contact lenses | | | | | |

### 7.2. Detailed Study Procedures

VISIT 1

Note that the subject must be wearing their habitual soft contact lenses into Visit 1.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |

| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
|---|---|---|
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Baseline<br>Questionnaires | The subject will respond to the following questionnaires: 1. CLUE Baseline Questionnaire 2. GSI Background Questionnaire |
| 1.7 | Other Questionnaires | The subject will respond to additional questionnaires: 1. Activity History |
| 1.8 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.9 | Remove Habitual<br>Lens | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. |
| 1.10 | Slit Lamp Findings | FDA Slit Lamp Classification Scale ( will be used to grade the findings and will be used to determine eligibility. Record only whole numbers. If any of these slit lamp findings are Grade 3 or higher, the subject is ineligible to continue but may return at a later date to complete another Baseline. If after a total of 2 attempts the subject is deemed ineligible, then complete the Final Evaluation. Limbal and Bulbar Conjunctival Hyperemia findings using the 0.5 increment scale, and Corneal Staining Assessment will be emphasized using the 1.0 |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | increment scale for internal purposes only. | |
| 1.11 | Iris Color | The investigator will record the subject's iris color based on the scale provided. | Appendix E |
| 1.12 | Subjective Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. Best corrected distance visual acuity (BVA) must be 20/25+3 or better in each eye. | |
| 1.13 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. | |
| 1.14 | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.15 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. |
| 1.16 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 1.17 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.18 | Subjective Best<br>Sphere Over<br>Refraction and<br>Modification | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.19 | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |
| 1.20 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.21 | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 1.22 | Distance ETDRS<br>logMAR Visual<br>Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 1 • The left eye will read Chart 2 |
| 1.23 | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 1.24 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Snellen visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 1.25 | Dispense | The lenses will be dispensed for 6-8 days 1. The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>per day, ≥5 days per week.</li> <li>2. The lenses will be worn as daily wear only.</li> <li>3. All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>4. Preservative-free rewetting drops are permitted if needed.</li> <li>5. A patient instruction booklet will be provided.</li> <li>6. The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> </ul> |

### VISIT 2

The follow-up will occur 6-8 days after the initial dispensing. The subjects must enter the visit wearing their study contact lenses.

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. |
| 2.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.5. | Preference | Subjects will respond to a preference questionnaire comparing study lens 1 to their habitual lenses. |

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 2.6. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance |
| 2.7. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.8. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 2.9. | Surface Deposits | Record any front and back surface lens deposits. |
| 2.10. | Temporary Lens<br>Removal & Storage | Both lenses will be removed and temporarily stored in a lens case with either saline or Optifree® Puremoist®. The lenses will be reinserted in step 2.13. |
| 2.11. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be Grade 2 or less as graded on the FDA scale continue onto Trial Period 2. If the subject is not eligible, they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors |

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| | | immediately. |
| 2.12. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. |
| 2.13. | Lens Reinsertion | The lenses removed in step 2.10 will be reinserted. The subject will wear the same lenses an additional 6-8 days to their next scheduled visit. |
| 2.14. | Exit Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |

### VISIT 3

The follow-up will occur 6-8 days following Visit 2. The subjects must enter the visit wearing their study contact lenses.

| Visit 3: Treatment 1 Follow-Up 2 | | | | | |
|---|---|---|--|--|--|
| Step | Procedure | Details | | | |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. | | | |
| 3.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | | | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. | | | |
| 3.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | | | |
| 3.5. | Preference | Subjects will respond to a preference questionnaire comparing study lens 1 to their habitual lenses. | | | |
| Visit 3: Treatment 1 Follow-Up 2 | | | |
|---|---|---|---|
| Step | Procedure | Details | CTP |
| 3.6. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | |
| 3.7. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 3.8. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 1 • The left eye will read Chart 2 | |
| 3.9. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories | |
| 3.10. | Surface Deposits | Record any front and back surface lens deposits. | |
| 3.11. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVC for 45 days after LSLV for laboratory testing (Section 7.4). | |
| 3.12. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar | |

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | CTP |
| | | Conjunctival Hyperemia findings<br>and Corneal Staining Assessment<br>will be emphasized using a more detailed<br>scale. | |
| | | Note: Findings must be grade 2 or less as graded on the FDA scale to continue onto Trial Period 2. If the subject is not eligible, they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. | |
| 3.13. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. | |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 3.14. | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. |
| 3.15. | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 3.16. | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 3.17. | Subjective Best<br>Sphere Over<br>Refraction | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. |
| 3.18. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 3.19. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 3.20. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 3.21. | Distance ETDRS<br>logMAR Visual<br>Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 3 • The left eye will read Chart 4 |
| 3.22. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 3.23. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 3.24. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free®</li> </ol> |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | PureMoist® to be used in a rub regime. 4. Preservative-free rewetting drops are permitted if needed. 5. The lenses must be stored in the supplied case out of direct sunlight. |
| | | Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit). |
| | | Note 2: The subject's habitual contact lenses cannot be worn at any time during the study. |

VISIT 4

The follow-up will occur 13-15 days after the dispensing of the second study lenses. The subjects must enter the visit wearing their study contact lenses.

| | Visit 4: Treatment 2 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. |
| 4.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 4.5. | Lens Preferences | Subjects will respond to the preference questionnaire comparing study lens 1 and study lens 2. |
| 4.6. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up |

| | Visit 4: Treatment 2 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| | | 2. GSI Product Performance |
| 4.7. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 4.8. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 1 • The left eye will read Chart 2 |
| 4.9. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 4.10. | Surface Deposits | Record any front and back surface lens deposits. |
| 4.11. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). |
| 4.12. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. |

| | Visit 4: Treatment 2 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| | | Note: Findings must be grade 2 or less as graded on the FDA scale to continue onto Trial Period 2. If the subject is not eligible, they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. |
| 4.13. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. |

| | Visit 4: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 4.14. | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. Record the test condition. |
| 4.15. | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 4.16. | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 4.17. | Subjective Best<br>Sphere Over<br>Refraction | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of $\pm 0.00$ D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. |
| 4.18. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |
| 4.19. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |

| | Visit 4: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 4.20. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 4.21. | Distance ETDRS<br>logMAR Visual<br>Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 3 • The left eye will read Chart 4 |
| 4.22. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 4.23. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 4.24. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime. </li> <li>Preservative-free rewetting drops are permitted if needed.</li> </ol> |

| | Visit 4: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | 5. The lenses must be stored in the supplied case out of direct sunlight. |
| | | Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit). |
| | | Note 2: The subject's habitual contact lenses cannot be worn at any time during the study. |

## VISIT 5

The follow-up will occur 13-15 days after the dispensing of the third study lenses. The subjects must enter the visit wearing their study contact lenses.

| | Visit 5: Treatment 2 Follow-Up | |
|---|---|---|
| Step | Procedure | Details |
| 5.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 5.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 5.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. |
| 5.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 5.5. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance |
| 5.6. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |

| Visit 5: Treatment 2 Follow-Up | | |
|---|---|---|
| Step | Procedure | Details |
| 5.7. | logMAR (ETDRS)<br>Visual Acuity | Perform 4 m distance ETDRS logMAR visual acuity test OD and OS under the following conditions: • Bright illumination (e.g., >400 lux), with high contrast charts (HLHC); • The right eye will read Chart 1 • The left eye will read Chart 2 |
| 5.8. | Subjective Lens Fit<br>Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 5.9. | Surface Deposits | Record any front and back surface lens deposits. |
| 5.10. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). |
| 5.11. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be Grade 2 or less as graded on the FDA scale Otherwise they must be followed as an adverse event. Adverse events must be reported to the JJVC monitors immediately. |

| Visit 5: Treatment 2 Follow-Up | | |
|---|---|---|
| Step | Procedure | Details |
| 5.12. | Eye Rinse | The study coordinator, investigator, or technician will rinse the subject's eyes thoroughly with saline. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |
| F.2 | Best-corrected Distance Visual Acuity Record the subject's best corrected distance visual acuity with refraction OD, OS, and OU. | |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

CR-5960, v2.0


JJVC CONFIDENTIAL

The following information will be collected during an unscheduled visit.

| Step | Procedure | Details |
|---|---|---|
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Change of Medical<br>History and Concomitant<br>Medications | Questions regarding the change of subjects' medical history and concomitant medications. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.4 | Subjective Sphero-<br>cylindrical Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. |
| U.5 | Slit Lamp Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If no slit lamp finding is noted on the EDC form it is considered as a zero "0" Grade for all observations listed. |
| | | After the slit lamp examination, at the discretion of the Investigator, rinse the subject's eyes thoroughly with preservative-free saline. |
| U.6 | Dispensing (if applicable) | Additional lenses may be dispensed if one is lost or torn during the wearing period. |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS and OU) to the nearest letter. |

# 7.4. Laboratory Procedures

The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

The disposition (accountability) of all enrolled subjects will be presented by study lens and overall to show the number and percentage of subjects in each of the following status subgroups:

- 1. Completed: Subjects are considered to have completed the study if they have completed all scheduled visits.
- 2. Discontinued: Subjects are considered to have discontinued from the study if they are (i) randomized (ii) Successfully Dispensed and (iii) discontinued because of one of the following reasons: a) Withdrew Consent (b) Lost to Follow Up (c) Subject no longer meets eligibility criteria (e.g. pregnancy) (d) Subject withdrawn by PI due to non-compliance to protocol (e) Discontinuation of study treatment as a result of the investigator's belief that for safety (f) Reasons it is in the best interest of the subject to stop treatment (g) Study lens no longer available (h) A scheduled visit was missed.
- 3. Total dispensed: Completed + Discontinued
- 4. Enrolled not Successfully Dispensed: Subjects are considered to be Enrolled Not Successfully Dispensed Subjects if they were (i) enrolled to the study (provided informed consent) but failed to satisfy the eligibility criteria (inclusion/exclusion criteria), (ii) were not randomized to study lens for any reason or (iii) if they are randomized but did not satisfactorily complete the dispensing process. This includes subjects who were dispensed a different type of study lens for each eye or who were dispensed same study lens for both eyes but did not return for any follow-up visits.
- 5. Total enrolled: Completed + Discontinued + Enrolled not Successfully Dispensed
- 6. The percentage will be calculated using total enrolled as denominator.
- 7. Safety and efficacy analysis sets will be defined as subsets of dispensed subjects (Completed + Discontinued).

### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol (e.g. Subject more than 2 days out of visit window).
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)

- Subject develops significant or serious adverse events causing discontinuation of study lens wear (subjects missing more than 2 days of missed lens wear within a period 1 of week should be discontinued)
- Subjects who have experienced a Corneal infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed any scheduled study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 0
- Collect all unused test article(s) from the subject

Investigator will discuss with sponsor before enrolling any additional subjects if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: See section 3.3

Concomitant therapies that are disallowed include: See section 3.3

### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented


deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)".
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.

• Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether or not the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eve Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (for test article return instructions)

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is any untoward (unwanted) medical occurrence in a patient or clinical investigation subject administered a test article, study treatment or study procedure

whether or not caused by the test article, study treatment or procedure. An AE can therefore be any unfavorable or unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of the test article, study treatment, or study procedure whether or not related to the test article, study treatment, or study procedure.

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

# **Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – A sub-set of AEs, and include only those adverse events that are cause by or related to the investigational device.

**Unanticipated Adverse Device Effect (UADE)** – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; doubtful; possible; probable; very likely see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2).
- Outcome Not Recovered or Not Resolved; Recovering or Resolving; Recovered or Resolved with Sequelae; Recovered or Resolved; Death Related to Adverse Event; Unknown
- Actions Taken None; temporarily discontinued; permanently discontinued; other action taken

#### 13.2.1 Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article, study treatment, or study procedure. The test article, study treatment or study procedure relationship for each adverse event shall be determined by the Investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2 Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities


• Severe – Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment /eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the test article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether or not a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event /eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether or not the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1 Reporting Adverse Events to Sponsor

### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article

• Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

### 13.4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.5. Event of Special Interest

None

### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the course of the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

### 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC).

## **Description of Summary Tables:**

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables for each subject/eye by study lens type (as appropriate). All variables will be summarized on the safety population. Analysis variables will be summarized on both the analysis and safety populations. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data. Unscheduled visits will be summarized separately if applicable.

### 14.2. Sample Size Justification

This study was designed and powered to show non-inferiority of the Test lens compared to the Control lens with respect to CLUE Comfort, logMAR Visual Acuity and Slit Lamp Findings (Grade 3 or higher). It was assumed there was no difference between the Test and Control lens with respect to CLUE comfort, visual performance and slit lamp findings.

In addition to the endpoints mentioned above this study was also powered to demonstrate the proportion of eyes with acceptable fitting on the Test lens is significantly superior to 90% as wells as the cumulative odds ratio of (individual reduction items) the Test lens compared to the control lens is significantly superior to 1.00.

Unless otherwise specified, the sample size was calculated to achieve a minimum statistical power of 80% and a type I error of 5%.

| The sample size calculation was based on | historical data from a four similar randomized |
|---|---|
| bilateral multi-site studies | where the same |
| Test and Control lenses were used. Both ler | nses were worn as daily wear for at least 5 days |
| 1 1 | ow-up visits occurred at 1 and 2-weeks after the |
| initial visit. Subject accountability for each s | study is listed in Table 4 below. |



Table 6: Descriptive Summary of Slit Lamp Findings Pooled Across Historical Studies



<sup>%=</sup> nx100/N; SD=Standard Deviation

# **CLUE Comfort**

Sample size calculation for CLUE comfort was carried out using an approximation of the power of an F-test derived from the non-centrality parameter calculated form the observed F statistic of a linear model<sup>8</sup>.

<sup>&</sup>lt;sup>1</sup>All SLF reported for this study are combined for the purposes of summarizing

<sup>&</sup>lt;sup>2</sup> The percent (%) of Any Grade 2 is calculated using the Total Unique Eyes as the denominator

### Model details:

CLUE comfort was analyzed using a linear mixed model. Lens type, period and the interaction between lens type and period were included in the model as fixed effects. A compound symmetric (CS) covariance was used to model the correlation between measurements on the same subject across study periods. Below is the variance-covariance matrix used in the CLUE Comfort model.

$$\sum_{comfort} \begin{pmatrix} 202 & 105 & 105 \\ 105 & 202 & 105 \\ 105 & 105 & 202 \end{pmatrix}$$

#### **Visual Performance**

The sample size calculation for distance monocular visual performance was performed assuming that there was no difference between the Test and Control lenses to achieve a minimum statistical power of 80%. Assuming a mean of 0 LogMAR, a standard deviation of 0.10 (based on historical ACUVUE® OASYS®) and a correlation between eye of 0.80, 2000 replicating trials were simulated for the repeated measurements from the multivariate normal distribution

### **Acceptable Lens Fit**

Acceptable lens fit is a binary response as y=1 if a subject eye has an acceptable fit and 0 otherwise. The common reference rate of 95% was selected for the sample size calculation, since this is considered to be a more conservative reference proportion. Assuming a correlation 0.80 between measurements within the same subject and period; and assuming a correlation of 0.50 between measurements within the same subject across periods. A total of 2000 replicating trials were simulated to estimate a sample size with a minimum statistical power of 80%.

#### **Slit Lamp Findings**

There was no Grade 3 or higher SLFs in any of the four historical studies. Therefore an incidence rate of 0.5% was chosen based on previous research literature<sup>3, 4</sup>. Assuming a correlation 0.50 between measurements within the same subject and period; and assuming a correlation of 0.30 between measurements within the same subject across periods. A total of 2000 replicating trials were simulated to estimate a sample size with a minimum statistical power of 80%.

Table 7: Sample Size Estimates and Power Calculations for Primary Endpoints

| Endpoint | Number per Subjects to Complete | Power |
|----------------------------------|---------------------------------|-------|
| Distance Monocular Visual Acuity | 40 | >99% |
| SLFs Grade 3 or Higher | 120 | 86% |
| Acceptable lens Fit | 70 | 83% |
| CLUE Comfort | 60 | 80% |


#### 14.3. Analysis Populations

A separate Statistical Analysis Plan (SAP) will be provided for this study. If there are any discrepancies between the protocol and the SAP, the SAP will supersede the statistical sections in the protocol.

## **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

# **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

The primary and secondary hypotheses will be tested with a type I error of 5% individually.

## 14.5. Primary Analysis

Primary efficacy analysis:

#### Visual Acuity

Distance monocular visual acuity (logMAR) will be analyzed using a Bayesian multivariate normal random-effects model to compare the Test and control lenses. The regression model will include sequence of lens wear, lens type and first-order carryover effect as fixed effects. Clinical site and subject nested within clinical site will be included as random effects. Other subject characteristics such as gender and age will be included as fixed effects when appropriate.

#### The Model:

Let  $y_{ijklm} = (y1_{ijklm}, y2_{ijklm}, y3_{ijklm})$  denote the visual acuity (logMAR) for the  $m^{th}$  subject at the  $l^{th}$  site, assigned to the  $i^{th}$  lens for the  $j^{th}$  eye using the  $k^{th}$  sequence at periods 1, 2, 3, respectively. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{ijklm} \sim N(\mu_{ijklm}, \Sigma)$$

Where  $\mu_{ijklm} = (\mu 1_{ijklm}$ ,  $\mu 2_{ijklm}$ ,  $\mu 3_{ijklm})^T$  and  $\Sigma$  is a 3X3 variance-covariance matrix. Here,

$$\begin{split} & \mu \mathbf{1}_{ijklm} = \mu_0 + \ \pi_1 + \beta_1 Lens_{i[j,k]} + \beta_4 Sequence_k + \\ & \mu \mathbf{2}_{ijklm} = \mu_0 + \ \pi_2 + \beta_2 Lens_{i[j,k]} - \ \beta_4 Sequence_k + \beta_5 Carry \mathbf{1}_{i[j,k]} + \gamma_l + \delta_{l_{(m)}} + \alpha_{j_{(m(l))}} \end{split}$$

$$\mu 3_{ijklm} = \mu_0 + \pi_3 + \beta_3 Lens_{i[j,k]} + \beta_4 Sequence_k - \beta_5 Carry 1_{i[j,k]} + \gamma_l + \delta_{l(m)} + \alpha_{j_{(m(l))}}$$

In this model  $\pi_1$ ,  $\pi_2$ ,  $\pi_3$  represent the effect of period with the constraint  $\pi_1 + \pi_2 + \pi_3 = 0$ . In Lens I will be determined by the subject eye j and sequence k, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the control lens and  $Lens_i=1$  for the Test lens, sequence is defined as: Sequence=0 for the order Control/Test/Test and Sequence=1 for order Test/Control/Control. The first-order carryover effect will be defined as carry=0 for the Control lens and carry=1 for the Test lens. So  $\beta_1$  stands for the difference between the Test and control lens with respect to visual performance at period 1. A negative  $\beta_2$  indicates the Test performed better than the control lens.

We assume random subject eye effects are independent and identically distributed (i.i.d) as  $\alpha_{j_{(m(l))}} \sim N(0, \sigma_{eye/subject/site}^2)$  as random eye nested within subject within clinical site, the random subject effect are i.i.d as  $\delta_{l_{(m)}} \sim (0, \sigma_{subject/site}^2)$  as random subject nested within clinical site and the random site effect is i.i.d as  $\gamma_l \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2 (sequence), carry1=1, 2 (first-order carryover effect) and l=1...|  $m_l$ (subject/site) and l=1,2,3,4 and 5 (site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effects  $\sigma^2_{eye/subject/site}$ ,  $\sigma^2_{subject/site}$  and  $\sigma^2_{site}$  independent non-informative conjugate priors inverse-gamma(0.001, 0.001) will be used. For  $\Sigma$ , non-informative conjugate priors inverse-wishart(3,S) will be used where S is a 3X3 variance-covariance matrix of  $y_{ijklm}$ . The metropolis sampler algorithm as implemented in the SAS/STAT MCMC procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

#### Hypothesis Testing

The null and alternative hypothesis for visual acuity (logMAR) to test for non-inferiority of the Test lens relative to the control lens is as follows:

$$H_o: \frac{\beta_1 + \beta_2 + \beta_3}{3} \ge 0.05$$
  
 $H_A: \frac{\beta_1 + \beta_2 + \beta_3}{3} < 0.05$ 

Non-inferiority will be declared if the upper limit of the 95% credible interval of the difference between the Test and Control is below 0.05, i.e.  $P(\frac{\beta_1+\beta_2+\beta_3}{3}<0.05)\geq 0.975$ . Superiority will be established if the upper limit of the 95% credible interval of the difference between the Test and Control lens is below 0.0, i.e.  $P(\frac{\beta_1+\beta_2+\beta_3}{3}<0.0)\geq 0.975$ . Superiority will be tested only if non-inferiority is met.

### **CLUE Overall Comfort**

CLUE Comfort scores will be analyzed using a Bayesian multivariate normal random-effects model to compare the Test and control lenses. The regression model will include baseline CLUE comfort scores, sequence of lens wear, lens type and first-order carryover as fixed


effects. Clinical site will be included as random effects. Other subject characteristics such as age, gender, race and iris category will be included when appropriate.

#### The Model:

Let  $y_{ijkl} = (y1_{ijkl}, y2_{ijkl}, y3_{ijkl})$  denote the CLUE Comfort score for the  $l^{th}$  subject at the  $k^{th}$  site, assigned to the  $i^{th}$  lens using the  $j^{th}$  sequence at periods 1, 2 and 3. The likelihood for  $y_{ijkl}$  is constructed as follows:

$$y_{iikl} \sim N(\mu_{iik}, \Sigma)$$

Where 
$$\mu_{ijkl} = (\mu 1_{ijkl}, \mu 2_{ijkl}, \mu 3_{ijkl})^T$$
 and  $\Sigma$  is a 3X3 variance-covariance matrix. Here,  $\mu 1_{ijkl} = \mu_0 + \pi_1 + \beta_1 Lens_{[i,j]} + \beta_4 baseline + \beta_5 Sequence_j + \gamma_k$   $\mu 2_{ijkl} = \mu_0 + \pi_2 + \beta_2 Lens_{[i,j]} + \beta_4 baseline - \beta_5 Sequence_j + \beta_6 Carry 1_{[i,j]} + \gamma_k$   $\mu 3_{ijkl} = \mu_0 + \pi_3 + \beta_3 Lens_{[i,j]} + \beta_4 baseline + \beta_5 Sequence_j - \beta_6 Carry 1_{[i,j]} + \gamma_k$ 

In this model  $\pi_1, \pi_2, \pi_3$  represent the effect of period with the constraint  $\pi_1 + \pi_2 + \pi_3 = 0$ . Lens I will be determined by sequence j, therefore i is denoted as a function of j. We define Lens=0 for the control lens and Lens = 1 for the Test lens, sequence is defined as: Sequence=0 for the order Control/Test/Test and Sequence=1 for order Test/Control/Control. The first-order carryover effect will be defined as carry=0 for the Control lens and carry=1 for the Test lens. So  $\beta_1$  stands for the difference between the Test and Control lens with respect to CLUE comfort; A positive  $\beta_1$  indicates the Test performed better than the control.

We assume random site effect is independent and identically distributed (i.i.d) as  $\gamma_k \sim N(0, \sigma_{site}^2)$  for site for i=1, 2 (lens), j=1, 2, (sequence), k=1,2, 3, 4 and 5 (site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effect of  $\sigma_{site}^2$  an independent non-informative conjugate prior, inverse-gamma(0.001, 0.001) will be used. For  $\Sigma$ , non-informative conjugate priors inverse-wishart(3,S) will be used where S is a 3X3 variance-covariance matrix of  $y_{ijkl}$ . Starting values for the mean and variance of CLUE scores will be 60 and 400 (since standard deviation of CLUE is normalized to be 20), respectively. The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

### **Hypothesis Testing**

The null and alternative hypotheses for CLUE comfort non-inferiority of the Test lens relative to the control lens are as follows:

$$H_o: \frac{\beta_1 + \beta_2 + \beta_3}{3} \leqslant -5$$

$$H_A: \frac{\beta_1 + \beta_2 + \beta_3}{3} > -5$$

Non-inferiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between the Test lens and the control lens is greater than -5, i.e.,  $P(\frac{\beta_1 + \beta_2 + \beta_3}{3} > -5) \ge 0.975$ . Superiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between the Test and Control lens is greater than 0, i.e.,  $P(\frac{\beta_1 + \beta_2 + \beta_3}{3} > 0) \ge 0.975$ . Superiority will only be tested if non-inferiority is established.

# **Lens Fit Acceptance**

Lens fit acceptance will be analyzed using a Bayesian Logistic regression random-effects model to estimate the proportion of subjects eyes wearing the Test lens having acceptable lens fitting. The regression model will include period, sequence of lens wear and first order carryover effect. Site, subject nested within site and eye within subject within site will be included in the model as random effects.

Let  $y_{ijklm}=1$  if an acceptable lens fit is observed for eyes wearing the Test lens only and  $y_{ijklm}=0$  otherwise for the  $m^{th}$  subject, from the  $l^{th}$  site, for the  $i^{th}$  eye in the  $j^{th}$  period using the  $k^{th}$  sequence.

$$y_{iiklm} \sim Binary (p_{iiklm})$$

$$p_{ijklm} = \frac{exp(\textit{Numerator})}{1 + exp(\textit{Numerator})}$$

 $\begin{aligned} Numerator &= \beta_0 + \beta_1 Lens_{i[j,k]} + \beta_3 period_{j1} + \beta_4 period_{j2} + \beta_5 sequence_k + \beta_6 Carry \mathbf{1}_{i[j,k]} + \gamma_1 + \delta_{m_{(l)}} + \alpha_{j_{(m(l))}} \end{aligned}$ 

We assume the random subject eye effects are i.i.d as  $\alpha_{j_{(m(l))}} \sim N(0, \sigma_{eye/subject/site}^2)$  for eye nested within subject within clinical site, the random effect for subject are i.i.d as  $\delta_{m_{(l)}} \sim N(0, \sigma_{subject/site}^2)$  for subject nested within clinical site and the random clinical site effects are i.i.d as  $\gamma_m \sim N(0, \sigma_{site}^2)$  for i=1, 2 (eye), j=1, 2, 3 (period) k=1, 2(Sequence) l=1, ...5 (Site) m=1, ... $n_l$ (subject/site).

For the  $\beta$  coefficients, independent non-informative priors N(0, 10000) will be used. For the variance of random effects of  $\sigma^2_{eye/subject/site}$ ,  $\sigma^2_{subject/site}$  and  $\sigma^2_{site}$ , independent non-informative conjugate priors inverse-gamma (0.001, 0.001) will be used. The Metropolis-Hastings algorithm as implemented in the SAS/STAT 14.1 PROC MCMC procedure will be used to estimate posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

# **Hypothesis Testing**

With respect to Acceptable lens fit the null and alternative hypothesis for superiority is as follows:

$$H_0 = p \le 0.90$$
  
 $H_1 = p > 0.90$ 


Where, p represents the proportion of subject eyes that achieve acceptable fit for the Test lens.

Success for acceptable fit will be declared if the lower bound of the 2-sided 95% credible interval of the proportion is greater than 0.90; i.e.  $P(P > 0.90) \ge .975$ .

Primary safety analysis:

# **Slit Lamp Findings**

Grade 3 or higher slit lamp findings will be analyzed using a Bayesian Logistic regression random-effects model to compare the Test and Control lenses. The regression model will include baseline slit lamp findings, lens type, period, sequence of lens wear and first order carryover effect. Site, subject nested within site and eye within subject within site will be included in the model as random effects.

Let  $y_{ijklmn}$ =1 if a Grade 3 or higher SLF is observed and  $y_{ijklm}$  =0 otherwise for the  $n^{th}$  subject, from the  $m^{th}$  site, assigned to the  $i^{th}$  study lens for the  $j^{th}$  eye in the  $k^{th}$  period using the  $l^{th}$  sequence.

$$y_{ijklmn} \sim Binary (p_{ijklmn})$$

$$p_{ijklmn} = \frac{exp(\textit{Numerator})}{1 + exp(\textit{Numerator})}$$

Numerator= 
$$\beta_0 + \beta_1 Lens_{ij[k,l]} + \beta_2 Baseline SLF_1 + \beta_3 period_{k1} + \beta_4 period_{k2} + \beta_5 sequence_k + \beta_6 Carry1_{i[k,l]} + \gamma_m + \delta_{n_{(m)}} + \alpha_{j_{(n(m))}}$$

We assume the random subject eye effects are i.i.d as  $\alpha_{j_{(n(m))}} \sim N(0, \sigma_{eye/subject/site}^2)$  for eye nested within subject within clinical site, the random effect for subject are i.i.d as  $\delta_{n_{(m)}} \sim N(0, \sigma_{subject/site}^2)$  for subject nested within clinical site and the random clinical site effects are i.i.d as  $\gamma_m \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2 (eye), k=1, 2, 3 (period) l=1, 2 (Sequence) m=1, ...5 (Site) m=1, ... $n_m$  (subject/site).

In this model, the lens I will be determined by the period k and sequence l, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the Control lens and  $Lens_i=1$  for the Test lens.

For the  $\beta$  coefficients, independent non-informative priors N(0, 10000) will be used. For the variance of random effects of  $\sigma^2_{eye/subject/site}$ ,  $\sigma^2_{subject/site}$  and  $\sigma^2_{site}$ , independent non-informative conjugate priors inverse-gamma (0.001, 0.001) will be used. The Metropolis-Hastings algorithm as implemented in the SAS/STAT 14.1 PROC MCMC procedure will be used to estimate posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

# **Hypothesis Testing**

The null and alternative hypothesis for Non-inferiority is as follows:

$$H_o$$
: p =  $(p_{Test} - p_{Control}) \ge 0.05$ 

$$H_A$$
: p =  $(p_{Test} - p_{Control}) < 0.05$ 

Where p represents the difference between the proportion of subject's eyes with Grade 3 or higher SLFs of the test group compare to the control group. Non-inferiority will be established if the upper limit of the 2-sided 95% credible interval is below 0.05, i.e.  $P(p=p_{Test}-p_{control} < 0.05 | y)=0.975$ .

In the event that the number of Grade 3 or higher SLFs is too small Grade 2 or higher SLFs will be analyzed and tested as described above.

#### 14.6. Secondary Analysis

Secondary efficacy analysis:

# CLUE Overall Quality of Vision and Handling

CLUE Overall Quality of Vision and Handling will be analyzed and test in the exact same manner as CLUE Overall Comfort.

Secondary safety analysis:

Not Applicable

#### 14.7. Other Exploratory Analyses

Other efficacy analysis:

### **Lens Preferences:**

Lens preference items listed below will be analyzed separately using Bayesian multinomial models for nominal data.



The regression models will include lens wearing sequence, age and gender as fixed covariates when appropriate. Investigational site will be included as random effect if the variation across sites is not negligible.

Let  $y_{ijkl} = (y_{ijkl}, y_{ijk2}, y_{ijk3}, y_{ijk4})$  denote subject lens preference for the  $i^{th}$  subject from the  $j^{th}$  site with regard to the  $k^{th}$  preference item. Possible values of  $y_{ijkl}$  are:  $y_{ijk1} = 1$  if the subject preferred the Test lens, 0 otherwise;  $y_{ijk2} = 1$  if the subject preferred the Control lens, 0 otherwise;  $y_{ijk3} = 1$  if the subject preferred both the Test and Control lenses, 0 otherwise and  $y_{ijk4} = 1$  if the subject preferred neither Test nor Control lenses, 0 otherwise. The likelihood of  $y_{ijk4}$  is constructed as follow:

CR-5960, v2.0


JJVC CONFIDENTIAL

$$\begin{split} &y_{ijkl} \sim Multinomial \; (p_{ijk1}, \, p_{ijk2}, \, p_{ijk3}, \, p_{ijk4}) \\ &p_{ijkl} \; = \theta_{ijkl} \; / \; \Sigma_{m\theta_{ijkl}} \\ &\log(\theta_{ijkl}) = \mu_{0kl} + \beta_{1k} Sequence_{ij} + \beta_{2k} Age_{ij} + \beta_{3k} Female_{ij} + \delta_{j}, \end{split}$$

where  $\mu_{0kl}$  are the intercepts with  $\mu_{0k4}$  set to 0,  $p_{ijkl} = P(Y_{ijkl} = 1)$  and  $\gamma_j \sim N(0, \sigma_s^2)$ . We will use independent vague N(0,1000) priors for the regression coefficients  $\mu_{0kl}$ .  $\beta_{1k}$ ,  $\beta_{2k}$  and  $\beta_{3k}$ , and IG(0.001, 0.001) for  $\sigma_s^2$ .

## Hypothesis Testing:

For each preference item, the null and alternative hypotheses for superiority are as follows: Ho:  $OR_k \le 1$  Ha:  $OR_k > 1$ ; where  $OR_k$  represents the odds ratio of comparing the Test lens to the Control lens with regard to item k. The odds ratio is calculated as:

$$OR_k = p_{.k1}(1-p_{.k2})/p_{.k2}(1-p_{.k1}),$$

where  $p_{.kl}$  is the mean estimate  $p_{ijkl}$  for k=1, ..., 5 and l=1, ..., 4.

For each item k, the superiority will be declared if the lower bound of the 2-sided 95% credible interval of  $OR_k$  is greater than 1:  $Pr(OR_k > 1 | y) \ge .975$ .

# **Outdoor Glare Reduction**

Outdoor Glare reduction consists of 4 individual questionnaire items.



All outdoor glare items are assessed using the same ordinal scale (1=Excellent ...5=Poor). Outdoor Glare reduction items will be analyzed separately using a Bayesian multinomial model for ordinal data adjusting for baseline. The regression model will include sequence of lens wear, lens type, period and first order carryover effect. Clinical site and subject nested within clinical site will be included as random effects. Other subject characteristics such as age, gender, race and iris category will be included when appropriate.

#### The Model:

Let  $y_{ijklm} = (y_{ijklm1}, y_{ijklm2}, y_{ijklm3}, y_{ijklm4}, y_{ijklm5})$  denote the rating for the  $m^{th}$  subject, from the  $l^{th}$  site, assigned to the  $i^{th}$  study lens in the  $j^{th}$  period using the  $k^{th}$  sequence. Possible values of  $y_{ijklm}$  are 1 if the subject rating of outdoor glare items are X and 0 otherwise (x=1 for Excellent and X=5 for Poor, respectively). The likelihood is constructed as follows:


$$y_{ijklm}$$
 Multinomial  $(P_{ijklm1}, P_{ijklm2}, P_{ijklm3}, P_{ijklm4}, P_{ijklm5})$ 

$$P_{ijklm1} = \gamma_{ijklm1}$$

$$P_{ijklmX} = \gamma_{ijklmX} - \gamma_{ijklm(X-1)} \ 2 \le n \le 4$$

$$P_{ijklm5} = 1 - \sum_{x=1,...4} P_{ijklmX}$$

$$\text{Logit}(\ \gamma_{ijklmX}\ ) = \ \theta_n \ + \ \beta_1 Lens_{i[j,k]} \ + \ \beta_2 Period_{j1} \ + \ \beta_3 Period_{j2} \ + \ \beta_4 Sequence_k \ + \ \beta_5 Carry_{i[j,k]} \ + \ \gamma_l \ + \delta_{m_{(l)}}$$

Where  $\theta_n$  is the intercept for levels n=1,2,3,4,  $P_{ijklm1} = \Pr(\gamma_{ijklm1} = 1)$  with respect to outdoor glare preference. We assume the random subject effects are independent identically distributed (i.i.d) as  $\delta_{m_{(l)}} \sim N(0, \sigma_{subject/site}^2)$  for subject m nested within clinical site l and the random clinical site effects are i.i.d as  $\gamma_l \sim N(0, \sigma_{site}^2)$  for i=1,2 (lens), j=1, 2, 3 (Period) k=1, 2(Sequence) l=1, ...5 (Site) m=1, ... $n_l$ (subject/site).

In this model, the lens I will be determined by the period j and sequence k, therefore i is denoted as a function of j and k. We define  $Lens_i=0$  for the Control lens and  $Lens_i=1$  for the Test lens. The odds ratio for having higher rating can be written as  $OR=e^{-\beta 1}$ .

Independent vague N(0, 1000) priors for the regression coefficients  $\beta_i$  i=1,...5. For  $\theta_n$ , we are considering the following priors

$$\begin{array}{c} \pi 0(\theta 1) \sim N(0,100) \\ \pi 0(\theta 2|\; \theta 1) \sim N(0,100) I(\theta {>} \theta 1) \\ \pi 0(\theta 3|\; \theta 2) \sim N(0,100) I(\theta {>} \theta 2) \\ \pi 0(\theta 4|\; \theta 3) \sim N(0,100) I(\theta {>} \theta 3) \end{array}$$

For the variance of random effects independent vague normal priors will also be used;  $\sigma_P^2 \sim \text{inverse-gamma}(0.001, 0.001)$  and  $\sigma_S^2 \sim \text{inverse-gamma}(0.001, 0.001)$ . The Metropolis sample algorithim as implemented in the SAS/Stat MCMC Procedure will be used to estimate the posterior distributions of the unknown parameters. Inferences will be made based on the posterior credible interval for the relevant parameters.

#### Hypothesis Testing

The null and alternative hypotheses for superiority are as follows:

$$H_o$$
  $OR \leq 1$   
 $H_A$   $OR > 1$ 

Where OR represent the odds ratio of having higher rating of the Test lens compared to the Control lens. Superiority will be declared if the lower bound of the 2-sided 95% credible confidence interval is above 1, i.e.  $P(OR=e^{-\beta 1}>1|y)=0.975$ .

### **Indoor Glare Reduction**

Indoor Glare reduction consists of 4 individual questionnaire items:



Each item will be analyzed individually and tested in the exact same manner as the Outdoor Glare Reduction Items described above.

## **Driving Measures**

Driving measure consists of two individual questionnaire items:



### Hypothesis Testing

The null and alternative hypotheses for superiority are as follows:

$$H_o$$
  $OR \le 0.67$   
 $H_A$   $OR > 0.67$ 

Where OR represent the odds ratio of having higher rating of the Test lens compared to the Control lens. Non-inferiority will be declared if the lower bound of the 2-sided 95% credible confidence interval is above 0.67, i.e.  $P(OR = e^{-\beta 1} > 0.67 | y) = 0.975$ . Superiority will be declared if the lower bound of the 2-sided 95% credible interval is above 1, i.e.  $P(OR = e^{-\beta 1} > 1 | y) = 0.975$ . Superiority will only be tested in the event that non-inferiority is established.

Other safety analysis: Not Applicable

#### 14.8. Interim Analysis

There will not be an interim analysis performed on this study.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The

SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 10 imputations.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Data Sources for this study include: If external Data is collected outside of EDC, enter vendor contact information in this section of the protocol and type of external data collected. Enter information for each external data source.

- Vendor Name:
- Vendor Address:
- Vendor Contact:
- Phone:
- Email:
- Type of Data collected:

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-

Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.
# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013 and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)

- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

# 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and Sponsor policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

# 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Data Protection Act of 1998 and other applicable personal data


protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential

# 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of

a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

# 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Investigator's Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

Case Report Forms will be completed in real time according to the study procedures specified in the study protocol. Case Report Forms should be completed and reviewed and signed as applicable by the Investigator within 3 days of visit completion. Data queries must be addressed with complete responses within 3 days of generation. JJVC reserves the right to withhold remuneration until these activities are addressed.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

# 21. PUBLICATION

This study will be registered on ClinicalTrials.gov.

# 22. REFERENCES

1. Wirth, R.J., et al., *Development of the Contact Lens User Experience: CLUE Scales.* Optom Vis Sci, 2016. 93(8): p. 801-8.



8. W, S.W., Generalized linear mixed models. 2012, Boca Raton: CRC Press.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)

# APPENDIX B: PATIENT INSTRUCTION GUIDE

Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including torics, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUVUE OASYS® for ASTIG-MATISM contact lenses are that you must determine the stability, repeatability and drift angle of the lens axis so that you can prescribe the correct lens axis for your

## A. How to Determine Lens Cylinder and Axis Orientation

### Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks about 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position - there is no "top" and "bottom" as in a prism-ballasted lens, You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.



You'll need a biomicroscope and a 1 mm or 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eve. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark, It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring). it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- . Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is
- . Having supplemental spectacles to wear over the monovision contact lenses

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eve with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to

### B. How to Determine the Final Lens Power

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the patient's refractive axis, it is not advisable to over-refract because of the difficulty in computing the resultant power. In fitting contact lenses, it is customary to prescribe the full power in the sphere. In the cylinder, however, any lens rotation is visually disturbing to the patient, so it's more practical to prescribe as weak a cylinder as possible. So, here is how to determine the final lens power.

### For the Sphere:

If sphere alone or combined sphere and cylinder Rx >+4.00D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx ≤± 4.00D. vertex compensation is not necessary.

Adjust the axis by the drift angle using LARS. Choose a cylinder that is ≤ 0.25D from the refractive cylinder.

# Example 1

Manifest (spectacle) refraction: O.D. -2.50 -1.25 x 180 20/20

O.S. -2.00 -1.00 x 180 20/20

Choose a diagnostic lens for each eye with an axis as close to 180° as possible. Place the lens on each eye and allow a minimum of 3 minutes for

for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot pass state drivers licensing requirements with monovision correction.

- Make use of proper illumination when carrying out visual tasks
- Monovision fitting success can be improved by the following suggestions: Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients
- Emphasize the benefits of clear near vision and straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUC-TION GUIDE for these lenses. Copies are available for download at www. acuvue.com.

# PATIENT MANAGEMENT

# Dispensing Visit

- PROVIDE THE PATIENT WITH A COPY OF THE PATIENT INSTRUCTION. GUIDE FOR THESE LENSES. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULE (DISPOSABLE OR FREQUENT
- Recommend an appropriate cleaning and disinfecting system and provide the patient with instructions regarding proper lens care. Chemical or hydrogen peroxide disinfection is recommended.
- · Schedule a follow-up examination.

## Follow-up Examinations

- . Follow-up care (necessary to ensure continued successful contact lens wear) should include routine periodic progress examinations, management of specific problems, if any, and a review with the patient of the wear schedule, lens replacement schedule, and proper lens care and handling procedures.
- Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):
- 1. One week from the initial lens dispensing to patient
- One month post-dispensing
- Every three to six months thereafter

it to equilibrate, based on the patient's initial response to the lens. If the lens has not vet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx Prescribed:

O.D. -2.50 -1.25 x 180 O.S. -2.00 -0.75 x 180

### Example 2

Manifest (spectacle) refraction O.D. -3.00 -1.00 x 90 20/20

O.S. -4.75 -2.00 x 90 20/20

Choose diagnostic lenses of -3.00 -0.75 x 90 for the right eye and -4.50 -1.75 x 90 for the left eye, the nearest lenses available to the spherical power and axis needed. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable. The orientation mark on the right lens rotates left from the 6 o'clock position by 10°.

The fitting indicates the following:

### Right Eve:

Compensate the 10° axis drift by adding it to the manifest refraction axis. Here is the Rx prescribed: O.D. -3.00 -0.75 x 100

The lens on the left eye shows good centration, movement and a consistent tendency for the mark to drift right by 10° from the 6 o'clock position following a forced blink. Since the manifest refraction called for a power of -4.75D, adjust for the vertex distance and reduce the sphere by 0.25D and prescribe the -1.75D cylinder. Compensate for the 10° axis drift by subtracting it from the manifest refraction.

Here is the Rx Prescribed:

O.S. -4.50 -1.75 x 80

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

NOTE: More frequent or additional follow-up visits may be recommended for

- Preferably, at the follow-up visits, lenses should be worn for at least six hours. If the lenses are being worn for continuous wear, the examination should be performed as early as possible on the morning following overnight wear.
- · Recommended Procedures for Follow-Up Visits:
- Solicit and record patient's symptoms, if any.
- 2. Measure visual acuity monocularly and binocularly at distance and near with the contact lenses.
- 3. Perform an over-refraction at distance and near to check for residual refractive error.
- 4. With the biomicroscope, judge the lens fitting characteristics (as described in the GENERAL FITTING GUIDELINES) and evaluate the lens surface for deposits and damage
- 5. Following lens removal, examine the cornea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
- The presence of vertical corneal striae in the posterior central cornea and/ or corneal neovascularization is indicative of excessive corneal edema.
- The presence of comeal staining and/or limbal-conjunctival hyperemia. can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear, and/or a poorly fitting lens.
- Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.
- 6. Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

## WEARING SCHEDULE

The wearing and replacement schedules should be determined by the Eye Care Professional, Regular checkups, as determined by the Eye Care Professional, are also extremely important For Daily Wear:

# Patients tend to overwear the lenses initially. The Eve Care Professional should

emphasize the importance of adhering to the initial maximum wearing schedule Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to

# MULTIFOCAL FITTING GUIDELINES

### A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with the ACUVUE OASYS® for PRESBYOPIA contact lenses. Wear may not be optimal for activities such as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- 2. driving automobiles (e.g., driving at night). Patients who cannot pass their state driver's license requirements with these lenses should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

These lenses are not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise.

These lenses are available in the following ADD powers:

- Lens "LOW" = "low" near ADD lens (Max +1.25 ADD) Lens "MID" = "medium" near ADD lens (Max +1.75 ADD)
- Lens "HGH" = "high" near ADD lens (Max +2.50 ADD)

### **B. Fitting Instructions**

- 1. Determine the following:
- Eye dominance (the methods described in MONOVISION FITTING GUIDE-LINES may be used)
- . Spherical equivalent distance prescription (vertex corrected if necessary and rounded to less minus if between powers)
- Near ADD

For Extended Wear

- 2. Select the initial trial lens as follows:
- For each eve select the trial lens distance power that is closest to the patient's distance spherical equivalent,

The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

It is recommended that the contact lens wearer first be evaluated on a daily wear schedule. If successful, then a gradual introduction of extended wear can be followed as determined by the prescribing Eve Care Professional.

These lenses have been approved for extended wear up to 6 nights/7 days of continuous wear. Not all patients can achieve the maximum wear time.

For Therapeutic lens wear, close supervision by the Eve Care Professional is necessary. These lenses can be worn for extended wear for up to 6 nights/7 days of continuous wear. The Eye Care Professional should determine the appropriate wearing time and provide specific instructions to the patient regarding lens care, insertion, and removal.

# REPLACEMENT SCHEDULE

# For Lenses Prescribed for Frequent Replacement:

When prescribed for daily wear (frequent replacement), it is recommended that the lenses be discarded and replaced with a new lens every 2 weeks. However, the Eve Care Professional is encouraged to determine an appropriate replacement schedule based upon the response of the patient.

### For Lenses Prescribed for Disposable Wear: When prescribed for disposable wear, the replacement schedule should be deter-

mined by the Eve Care Professional based upon the patient's history and their ocular examination, as well as the practitioner's experience and clinical judgment. Once removed, it is recommended that the lens remain out of the eye for a period

of rest of overnight or longer and be discarded in accordance with the prescribed wearing schedule. The Eve Care Professional should examine the patient during the early stages of extended wear.


### · Select the near power of the lens based on the patient's ADD range as MONOVISION FITTING GUIDELINES

ADD: +0.75 to +1.25 use a "LOW" near ADD lens on each eye

ADD: +1.50 to +1.75 use a "MID" near ADD lens on each eve

ADD: +2.00 to +2.50 use a "HGH" near ADD lens on each eye

. Demonstrate the vision under various lighting conditions (normal and de-

. Make adjustments in power as necessary (see Multifocal Troubleshooting

• If distance and near vision are acceptable, perform a slit lamp examination to

dispensing and follow-up information in PATIENT MANAGEMENT).

Determine the amount of additional plus, or less minus, over one or both eves

vision is still not acceptable, change the non-dominant eye to the next highest

Determine the amount of additional minus, or less plus, over one or both eves

vision is still not acceptable, change the dominant eve to the next lowest ADD

that is acceptable while checking the effect on distance and near vision. If

power. If the patient is wearing two low ADD lenses, change the dominant

eye to a sphere lens with a power equal to the spherical equivalent distance

Determine the amount of additional plus and/or minus over one or both eyes

additional plus and/or minus is not required, change the lens power in the dom-

inant eye to the next lowest ADD power and the lens power in the non-domi-

that is acceptable while checking the effect on distance and near vision. If

All patients should be supplied with a copy of the PATIENT INSTRUCTION

LENS CARE DIRECTIONS

When lenses are dispensed, the Eye Care Professional should provide the patient

with appropriate and adequate warnings and instructions in accordance with the

should recommend an appropriate care system tailored to the patient's individual

For complete information concerning contact lens handling, care, cleaning, disin-

The Eve Care Professional should review with the patient, lens care directions for

cleaning, disinfecting and storing, including both basic lens care information and

The Eye Care Professional should review with patients that no cleaning or disinfec-

tion is needed with disposable lenses. Patients should always dispose of lenses

Lenses should only be cleaned, rinsed, and disinfected on an emergency basis

If the frequent replacement lens is off the eve and exposed to air from 30 minutes

to 1 hour or more, its surface will become dry and gradually become non-wetting. If

If the lens sticks (stops moving), the patient should be instructed to apply a

few drops of the recommended lubricating or rewetting solution directly to the

eye and wait until the lens begins to move freely on the eye before removing it.

If non-movement of the lens continues after a few minutes, the patient should

**EMERGENCIES** 

The patient should be informed that if chemicals of any kind (household products

gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the pa-

tient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY

CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY

when they are removed and have replacement lenses or spectacles available

specific instructions on the lens care regimen recommended for the patient.

fecting and storage, refer to the Patient Instruction Guide for these lenses. Copies

individual patient's lens type and wearing schedule. The Eve Care Professional

that is acceptable, while checking the effect on distance and near vision. If

assess adequate fit (centration and movement). If fit is acceptable, dispense

the lenses instructing the patient to return in one week for reassessment (see

Assess distance and near vision binocularly and monocularly.

creased illumination) and at distance, intermediate and near.

below). The use of hand-held trial lenses is recommended.

3. Allow the lens to settle for a minimum 10 minutes.

C. Multifocal Troubleshooting

Unacceptable Near Vision:

Unacceptable Distance Vision:

Unacceptable Distance and Near Vision:

are available for download at www.acuvue.com.

For Lenses Prescribed for Disposable Wear:

Care for a Dried Out (Dehydrated) Lens

Care for Sticking (Non-Moving) Lenses

immediately contact the Eye Care Professional.

ROOM WITHOUT DELAY

For Lenses Prescribed for Frequent Replacement Wear

when replacement lenses or spectacles are not available.

this should occur, discard the lens and use a new one.

nant eye to the next highest ADD power, if applicable.

GUIDE for these lenses. Copies are available for download at

prescription

www.acuvue.com.

### A. Patient Selection

### Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be deter mined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such

- 1. visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- 2. driving automobiles (e.g., driving at night). Patients who cannot pass their state driver's license requirements with monovision correction should be advised to not drive with this correction. OR may require that additional over-correction be prescribed.

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives. can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.

# B. Eve Selection

Generally, the non-dominant eye is corrected for near vision. The following two methods for eve dominance can be used.

# 1. Ocular Preference Determination Methods

lot number, and expiration date

Method 1: Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye

# HOW SUPPLIED

Each sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. The plastic package is marked with the • ACUVUE OASYSo: base curve, power, diameter, lot number, and expiration

- . ACUVUE OASYS for ASTIGMATISM: base curve, power, diameter,
- cylinder, axis, lot number, and expiration date ACUVUE OASYS® for PRESBYOPIA: base curve, power, diameter, ADD,

# REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with the lenses should be reported to:

> Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com



CJohnson & Johnson Vision Care Companies 2015 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc. Revision date: 06/15 Revision number: AO-06-15-01

> ACUMUE OASYS® and HYDRACLEAR® are trademarks of Johnson & Johnson Vision Care Companies

Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eve.

myopic) eye for distance and the more myopic (less hyperopic) eye for near.

3. Visual Demands Method Consider the patient's occupation during the eye selection process to deter-

best with the near lens on the left eye.

# 1. Unilateral Lens Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may only require a distance lens.

Example: A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without a lens. A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

# 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection in this Package Insert.

determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

IMPORTANT: Please read carefully and keep this

This Package Insert and Fitting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



ACUVUE OASYS® Brand Contact Lenses for ASTIGMATISM

ACUVUE OASYS® Brand Contact Lenses for PRESBYOPIA



sale by or on the order of a licensed practitioner.

for Daily and Extended Wear

CAUTION: U.S. Federal law restricts this device to

Other methods include the refractive error method and the visual demands

2. Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less

mine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

C. Special Fitting Characteristics

3. Trial Lens Fitting

Case history and standard clinical evaluation procedure should be used to

information for future use.

ACUVUE OASYS® Brand Contact Lenses

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker

Example: A secretary who places copy to the left side of the desk will function

## SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | DEFINITION |
|---|---|
| | Consult Instructions for Use |
| | Manufactured by or in |
| | Date of Manufacture |
| ₹ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterile Using Steam or Dry Heat |
| DIA | Diameter |
| BC | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| MAX ADD | Near ADD |
| LOW | "Low" Near ADD |
| MID | "Medium" Near ADD |
| HGH | "High" Near ADD |
| C€<br>0086 | Quality System Certification Symbol |
| Warecones | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| <b>R</b> Only | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| <u> </u> | Lens Orientation Correct |
| × | Lens Orientation Incorrect (Lens Inside Out) |

\*Topping-Off" is the addition of fresh solution to solution that has been sitting the case.

### Discard Date on Multi-Purpose Solution Bottle Instructions for Use

### Discard any remaining solution after the recommended time period indicated. on the bottle of multi-purpose solution used for disinfecting and scaking the contact lenses.

- The Discard Date refers to the time that the patient can safely use contact lens care product after the bottle has been opened. It is not the same as the expiration date, which is the last date that the product is still effective before it is opened.

### WARNING:

Using multi-numose solution beyond the discard date could result in contamination of the solution and can lead to severe infection, vision loss, or blindness.

- To avoid contamination, DO NOT touch tip of container to any surface. Replace cap after using.
- To avoid contaminating the solution, DO NOT transfer to other bottles or

### Rub and Rinse Time

### Instructions for Use

To adequately disinfect the lenses, the patient should rub and rinse the lenses according to the recommended lens rubbing and rinsing times in the labeling of the multi-purpose solution

### WARNING

- Rub and rinse lenses for the recommended amount of time to help prevent serious eve infections
- Never use water, saline solution, or rewetting drops to disinfect the lenses. These solutions will not disinfect the lenses. Not using the recommended disinfectant can lead to severe infection, vision loss, or blindness.

### Lens Case Care

- Empty and clean contact lens cases with digital rubbing using fresh, sterile disinfecting solutions/contact lens cleaner. Never use water. Cleaning should be followed by rinsing with fresh, sterile disinfecting solutions (never use water) and wiping the lens cases with fresh, clean tissue is recommended. Never air dry or recap the lens case lids after use without any additional cleaning methods. If air drying, be sure that no residual solution remains in the case before allowing it to air dry.
- Replace the lens case according to the directions provided by the Eye Care Professional or the manufacturer's labeling that accompanies the case.

### DESCRIPTION

The ACUVUE OASYS® Brand Contact Lenses, the ACUVUE OASYS® Brand Contact Lenses for ASTIGMATISM, and the ACUVUE OASYS® Brand Contact Lenses for PRESBYOPIA are soft (hydrophilic) contact lenses available as spherical, toric. or multifocal lenses and include HYDRACL FAR® PLUS Technology. The lenses are made of a silicone hydrogel material containing an internal wetting agent with visibility tinted UV absorbing monomer.

These lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. A benzotriazole UV absorbing monomer is used to block UV

The transmittance characteristics are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

| Lens Properties: | |
|---|---|
| <ul> <li>Specific Gravity (calculated):</li> </ul> | 0.98 – 1.12 |
| <ul> <li>Refractive Index:</li> </ul> | 1.42 |
| <ul> <li>Light Transmittance:</li> </ul> | 85% minimum |
| <ul> <li>Surface Character:</li> </ul> | Hydrophilic |
| <ul> <li>Water Content:</li> </ul> | 38% |
| <ul> <li>Oxygen Permeability:</li> </ul> | |
| VALUE | METHOD |
| 103 x 10 ¹¹ (cm²/sec)<br>(ml O₂/ml x mm Hg) @ 35°C | Fatt (boundary corrected, edge correct |
| 122 x 10 <sup>11</sup> (cm²/sec)<br>(ml O <sub>2</sub> /ml x mm Hg) @ 35°C | Fatt (boundary corrected, non-edge corrected) |

# Lens Parameters:

| Lens Faranieters. | |
|---|---|
| Diameter Range: | 12.0 mm to 15.0 mm |
| <ul> <li>Center Thickness:</li> </ul> | varies with power |
| <ul> <li>Base Curve Range:</li> </ul> | 7.85 mm to 10.00 mm |
| Spherical Power Range: | Daily Wear: -20.00D to +20.00D<br>Extended Wear: -20.00D to +14.00D |
| <ul> <li>Multifocal ADD Power Range:</li> </ul> | +0.25D to +4.00D |
| <ul> <li>Cylinder Power Range:</li> </ul> | -0.25D to -10.00D |

- Contact lens cases can be a source of bacterial growth.

# WARNING:

Axis Range:

Do not store lenses or rinse lens cases with water or any non-sterile solution. Only fresh multi-purpose solution should be used to prevent contamination of the lenses or lens case. Use of non-sterile solution can lead to severe infection, vision loss, or blindness.

2.5° to 180°

### **PRECAUTIONS**

### Special Precautions for Eve Care Professionals:

. Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient,
- Fluorescein, a vellow dve, should not be used while the lenses are on the eyes. The lenses absorb this dve and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eve use.
- . Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

### Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions:

### Handling Precautions

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- . DO NOT use if the sterile blister package is opened or damaged.
- · Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It

## **AVAILABLE LENS PARAMETERS**

The ACUVUE OASYS® Brand Contact Lenses are hemispherical shells of the following dimensions

14.0 mm

Center Thickness: Minus Lens - varies with power (e.g. -4.00D: 0.070 mm) Plus Lens - varies with power (e.g. +4.00D; 0.168 mm) Base Curve 8.4 mm, 8.8 mm

+6.50D to +8.00D (in 0.50D increments)

-0.50D to -6.00D (in 0.25D increments) -6.50D to -12.00D (in 0.50D increments) ±0.50D to ±6.00D (in 0.25D increments)

The ACUVUE OASYS® Brand Contact Lenses for ASTIGMATISM are hemitoric shells of the following dimensions:

Diameter:

Center Thickness: Minus Lens - varies with power (e.g. -4.00D: 0.080 mm) Plus Lens - varies with power (e.g. +4.00D: 0.172 mm)

Base Curve: 8.6 mm

> plane to -6.00D (in 0.25D increments) -6.50D to -9.00D (in 0.50D increments) +0.25D to +6.00D (in 0.25D increments)

Cylinder: -0.75D, -1.25D, -1.75D, -2.25D, -2.75D Axis: 10° to 180° (in 10° increments)

The ACUVUE OASYS® Brand Contact Lenses for PRESBYOPIA are hemispherical shells of the following dimensions:

Diameter:

Center Thickness: Minus Lens - varies with power (e.g. -4.00D: 0.070 mm) Plus Lens - varies with power (e.g. +4.00D: 0.168 mm)

Base Curve 9.4 mm Powers:

-9.00D to +6.00D (in 0.25D increments) ADD Powers: +1.25 (LOW), +1.75 (MID), +2.50 (HGH

> is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.

- . DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient Instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens contained unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container
- Do not touch the lens with fingernails
- · Close supervision is necessary for the Therapeutic use of these lenses. Ocular medications used during treatment with a bandage lens should be closely monitored by the Eye Care Professional. In certain ocular conditions, only the Eye Care Professional will insert and remove the lenses. In these cases, patients should be instructed not to handle the lenses themselves.

# Lens Wearing Precautions:

- . If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for Sticking (Non-Moving) Lenses". The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- . Never wear lenses beyond the period recommended by the Eve Care Professional.
- . The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.

# Lens Care Precautions:

- Different solutions cannot always be used together and not all solutions are safe for use with all lenses. Use only recommended solutions.
- Never use solutions recommended for conventional hard contact lenses
- Chemical disinfection solutions should not be used with heat unless

# TRANSMITTANCE CURVE

ACUVUE OASYS® Brand Contact Lenses vs. 24 yr. old human comea vs. 25 yr. old human crystalline lens



"The data was obtained from measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-1.00D lens, 0.070 mm center thickness). Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p.58, figure 2-21
 Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida,

1986, p.19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing evewear as directed.

# ACTIONS

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina. When hydrated and placed on the cornea for therapeutic use, the contact lens acts as a bandage to protect the

The transmittance characteristics are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation.

specifically indicated on product labeling for use in both heat and chemical

- Always use fresh, unexpired lens care solutions and lenses.
- Do not change solution without consulting with your Eve Care Professional.
- . Always follow directions in the package inserts for the use of contact lens
- Use only a chemical (not heat) lens care system. Use of a heat (thermal) care system can damage these lenses. Sterile unpreserved solutions, when used, should be discarded after the
- time specified in the directions. . Do not use saliva or anything other than the recommended solutions for lubricating or wetting lenses
- Always keep the lenses completely immersed in the recommended storage solution when the lenses are not being worn (stored). Prolonged periods of drying will reduce the ability of the lens surface to return to a wettable state. Follow the lens care directions in "Care For A Dried Out (Dehydrated) Lens' if lens surface does become dried out.

## Other Topics to Discuss with Patients:

- . Always contact the Eye Care Professional before using any medicine in the
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lens wear while such medication is being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned As with any contact lens, follow-up visits are necessary to assure the con-
- tinuing health of the patient's eves. The patient should be instructed as to a recommended follow-up schedule

# Who Should Know That the Patient is Wearing Contact Lenses?

the patient not wear contact lenses.

 Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.  Patients should always inform their employer of being a contact lens wearer.

Some jobs may require use of eye protection equipment or may require that

INDICATIONS (USES) The ACUVUE OASYS® Brand Contact Lens is indicated for the optical correction periods.

of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who have 1.00D or less of astigmatism. The ACUVUE OASYS® Brand Contact Lens for ASTIGMATISM is indicated for the

lowever, clinical studies have not been done to demonstrate that wearing

UV-Blocking contact lenses reduces the risk of developing cataracts or

other eye disorders. The Eye Care Professional should be consulted for

more information

UV radiation to the cornea and into the eve.

optical correction of visual acuity in phakic or aphakic persons with non-diseased eyes that are hyperopic or myopic and may have 10.00D or less of astigmatism. The ACUVUE OASYS® Brand Contact Lens for PRESBYOPIA is indicated for the optical correction of distance and near vision in presbyopic, phakic or aphakic persons with non-diseased eyes who may have 0.75D or less of astigmatism. These lenses contain a UV Blocker to help protect against transmission of harmful

Eve Care Professionals may prescribe the lenses either for single-use disposable wear or frequent/planned replacement wear with cleaning, disinfection and scheduled replacement (see "REPLACEMENT SCHEDULE"). When prescribed for frequent/planned replacement wear, the lenses may be cleaned and disinfected using a chemical disinfection system only.

These lenses have been approved for daily and extended wear for up to 6 nights/7 days of continuous wear, It is recommended that the contact lens wearer first be evaluated on a daily wear schedule. If successful, then a gradual introduction of extended wear can be followed as determined by the prescribing Eye Care Professional.

These lenses are also indicated for therapeutic use as a bandage lens for the following acute and chronic ocular conditions:

- · For corneal protection in lid and corneal abnormalities such as entropion, trichiasis, tarsal scars, and recurrent corneal erosion, In addition, they are indicated for protection where sutures or ocular structure malformation. degeneration or paralysis may result in the need to protect the cornea from exposure or repeated irritation.
- For corneal pain relief in conditions such as bullous keratopathy, epithelial. erosion and abrasion, filamentary keratitis, and post-keratoplasty.
- For use as a barrier during the healing process of epithelial defects such as chronic epithelial defects, corneal ulcer, neurotrophic and neuroparalytic keratitis, and chemical burns.
- For post surgical conditions where bandage lens use is indicated such as post refractive surgery, lamellar grafts, corneal flaps, and additional ocular

### ADVERSE REACTIONS

The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- . There may be a feeling of something in the eye (foreign body, scratched
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, and corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- . There may be excessive watering, unusual eye secretions or redness of the eve.
- . Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time
- . The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:
- How do the lenses feel on my eyes? How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATE-LY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL

If after inserting the new lens, the problem continues, the nationt should be

The patient should be instructed NOT to use a new lens as self-treatment for the The patient should be advised that when any of the above symptoms occur, a

serious condition such as infection, corneal ulcer, neovascularization or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

surgical conditions.

. For structural stability and protection in piggy back lens fitting where the cornea and associated surfaces are too irregular to allow for comeal rigid gas permeable (RGP) lenses to be fit. In addition, the use of the lens can prevent irritation and abrasions in conditions where there are elevation differences in the host/graph junction or scar tissue.

Lenses prescribed for therapeutic use may be worn for daily or extended wearing

## CONTRAINDICATIONS (REASONS NOT TO USE)

When prescribing contact lens wear for REFRACTIVE AMETROPIA USE, DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the
- . Any eye disease, injury or abnormality that affects the comea, conjunctiva or evelids
- · Severe insufficiency of lacrimal secretion (dry eye) Corneal hypoesthesia (reduced corneal sensitivity)
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses
- . Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.

Thimerosal, etc.) to which some people may develop an allergic response

- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (i.e., cleaning and disinfecting solutions, rewetting drops, etc.) that contain chemicals or preservatives (such as mercury or
- · Any active corneal infection (bacterial, fungal, protozoal or viral)
- If eves become red or irritated

For THERAPEUTIC USE, the Eye Care Professional may prescribe these lenses to aid in the healing process of certain ocular conditions, which may include those cited above.

# WARNINGS

Patients should be advised of the following warnings pertaining to contact

EYE PROBLEMS. INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

- Eye Discomfort
- Excessive Tearing.

## **GENERAL FITTING GUIDELINES**

### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses · Ability to follow instructions regarding lens wear care
- General health
- Ability to adequately handle and care for the lenses · Ability to understand the risk and benefits of lens wear

Patients who do not meet the above criteria should not be provided with

### contact lenses. B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the appropriate lens fitting instruction outlined below.

# C. Initial Power Determination

A spectacle refraction should be performed to establish the natient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D.

### D. Base Curve Selection (Trial Lens Fitting) The following trial lenses should be selected for patients regardless of keratome-

try readings. However, comeal curvature measurements should be performed to establish the patient's baseline ocular status.

- ACUVUE OASYS®: 8.4 mm/14.0 mm
- ACUVUE OASYS® for ASTIGMATISM: 8.6 mm/14.5 mm ACUVUE OASYS® for PRESBYOPIA: 8.4 mm/14.3 mm

The trial lenses should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

 Vision Changes, · Loss of Vision,

- Eve Redness.

### Or Other Eve Problems THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL

- When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious adverse reactions is increased when lenses are worn overnight, and that the risk of ulcerative keratitis is greater for extended wear contact lens users than for
- daily wear users.3 · Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- · Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products, including lens cases, are essential for the safe use of these products
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care, including cleaning the lens case.

<sup>a</sup>New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

Specific Instructions for Use and Warnings:

### Water Activity

Instructions for Use

Do not expose contact lenses to water while wearing them.

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

# Soaking and Storing Your Lenses

Instructions for Use Use only fresh multi-purpose (contact lens disinfecting) solution each time the

or blindness

lenses are soaked (stored) WARNING. Do not reuse or "top off" old solution left in the lens case since solution reuse reduces effective lens disinfection and could lead to severe infection, vision loss,

1. Criteria of a Properly Fit Lens A properly fit lens will center and completely cover the comea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered

# position when released.

2. Criteria of a Flat Fitting Lens A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete comeal coverage (i.e., limbal exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be flat

fitting, it should not be dispensed to the patient.

Criteria of a Steep Fitting Lens A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

### E. Final Lens Power (Spherical) A spherical over-refraction should be performed to determine the final lens

power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism. Example 1

| Diagnostic lens: | -2.00D |
|----------------------------|--------|
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | |

Diagnostic lens: -2.00D +0.25D Spherical over-refraction: -1.75D Final lens power:

# APPENDIX D: CLINICAL TECHNICAL PROCEDURES

Limbal and Conjunctival (Bulbar) Redness

**Expanded Sodium Fluorescein Corneal Staining** 

**Lens Fitting Characteristics** 

Subject Reported Ocular Symptoms/Problems

Front and Back Surface Lens Deposit Grading Procedure

Determination of Distance Spherocylindrical Refractions

Biomicroscopy Scale

Distance and Near Visual Acuity Evaluation

Distance logMAR Visual Acuity Measurement Procedure


# LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS
## EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING

### LENS FITTING CHARACTERISTICS

### SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS

## FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE

# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS

### BIOMICROSCOPY SCALE

#### DISTANCE AND NEAR VISUAL ACUITY EVALUATION

# DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

#### APPENDIX E: IRIS COLOR



#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: <u>CR-5960</u>, <u>Evaluation of Approved and Investigational Contact</u> Lenses

Version and Date: v2.0, 14 June 2017

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to GCP and ICH guidelines, the Declaration of Helsinki, ISO 14155, United States (US) Code of Federal Regulations (CFR), and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | Institution/Site Name | |
| | ilistitution/site ivame | |
| | Institution/Site Address | |

## **Electronic Signature Report**

Job Name: VIS-CR-005960/A-R&D Clinical Study Revision: VIS-CSPR-005796/2-Clinical Protocol Title: VIS Clinical Study Protocol Approval

Status: Approved

System: Vision Care R&D Knowledge Management

Generated By: Cook, Kara

Generated On: 2017-06-19 08:36:56

#### **Signoff Details**

| Function/Role | Approval Details | | |
|-------------------|------------------|----------|---------------------|
| Clinical Research | Participant | Decision | Decision Date |
| Manager | | Approved | 2017-06-15T11:18:35 |
| Approval | | | |

| Function/Role | | Approval Details | |
|---------------|-------------|------------------|---------------------|
| Clinician | Participant | Decision | Decision Date |
| Approval | | Approved | 2017-06-15T18:43:20 |

| Function/Role | | Approval Details | |
|-----------------|-------------|------------------|---------------------|
| Biostatistician | Participant | Decision | Decision Date |
| Approval | | Approved | 2017-06-15T16:07:34 |

